CLINICAL TRIAL: NCT05121584
Title: Evaluation of Two Different Types of Zirconia Crowns Used in Carious Primary Anterior Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arig Samir Abdelmonem Shawky (Other)
Responsible Party: Sponsor-Investigator, Arig Samir Abdelmonem Shawky, B.D.S, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pediatric Dentistry
Record Dates: First submitted 2021-11-14; First posted 2021-11-16 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Dental Caries in Children
Keywords: Zirconia crowns in pediatric dentistry; Dental caries; Aesthetic primary teeth restoration
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinder Krown (Experimental): Anterior primary teeth which restored by a Kinder Krown zirconia crown as a final restoration
  Interventions: Procedure: Placement of an anterior crown restoration as a final restoration
- NuSmile (Active Comparator): Anterior primary teeth which restored by a NuSmile zirconia crown as a final restoration
  Interventions: Procedure: Placement of an anterior crown restoration as a final restoration

INTERVENTIONS:
Procedure: Placement of an anterior crown restoration as a final restoration — Placement of an anterior crown restoration as a final restoration

SUMMARY:
Evaluation of two different types of zirconia crowns ( Kinder Krown , Nusmile crown) used in carious primary anterior teeth

DETAILED DESCRIPTION:
Assess the clinical and radiographic evaluation of Kinder Krowns and Nusmile crowns in restoring carious primary canines And compare between the two crowns used

ELIGIBILITY:
Inclusion Criteria:

* Children age ranging from 7 to 10 years
* Deep carious primary upper canines
* The tooth need pulpal treatment
* The tooth need a crown restoration
* The tooth not submerged
* The tooth is not mobile

Exclusion Criteria:

* Children with bruxism or deep bite
* Children with especial need
* Presence of pathological root resorption in preoperative x-ray
* Presence of tooth wear (abrasion/attrition) on the opposing teeth

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2022-03-21 (Estimated)

PRIMARY OUTCOMES:
Crown retention | 12 months
  Change in the following clinical assessment measure between baseline and 12 months using the scale below A=Intact B=Chipped/small but noticeable areas of loss of material C=Large loss of material D=Complete loss of crown
Opposing tooth wear | 12 months
  Binary (Yes/No)
Gingival health | 12 months
  Change in the following clinical assessment measure between baseline and 12 months using the scale below A=No inflammation B=Mild inflammation C=Moderate inflammation D=Marked inflammation
Immediate color match | 12 months
  A=No noticeable difference from adjacent teeth B=Slight shade mismatch C=Obvious shade mismatch
Gingival index (Loe and Silness) | 12 months
  Change in the following clinical assessment measure between baseline and 12 months using the scale below 0=Normal gingiva(natural colour pink gingiva no inflammation) 1=Mild inflammation(slight changes in colour,slight edema,no bleeding on probing) 2=Moderate inflammation(redness, edema and glazing, bleeding upon probing 3=Severe inflammation(marked redness and edema/ulceration/tendency to bleed spontaneously
Crown margins | 12 months
  Change in the following clinical assessment measure between baseline and 12 months using the scale below A=Continuous with the contour of the crown, nice adaptation B=Slight overhang or under contour present C=Large defects noted D=Restoration missing
Child/parent satisfaction | 12 months
  Binary(Yes/No)
Pathological external/internal root resorption | 12 months
  Binary(Present/Absent)
Periapical radiolucency | 12 months
  Binary(Present/Absent)

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Abdelmonem Elhendawy, Professor, Study Director — Tanta University; Fatma Ahmed Elshehaby, Professor, Study Director — Cairo University; Fatma Korany Ismail, Ass.Professor, Study Director — Cairo University; arig samir abdelmonem, bachelor, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No